CLINICAL TRIAL: NCT02165839
Title: Brief Behavioral Intervention for Insomnia During Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Oxana Palesh, Oxana Palesh PhD, MPH, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-30470; BRS0042 (Other: OnCore); 1R01CA181659-01A1 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-06-18 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Insomnia
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Eating Education Learning (HEAL) (Active Comparator): Control group.
  Interventions: Behavioral: Healthy Eating Education Learning (HEAL)
- Brief Behavioral Therapy for Insomnia (BBT-I) (Experimental)
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia (BBT-I)

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy for Insomnia (BBT-I)
  Arms: Brief Behavioral Therapy for Insomnia (BBT-I)
Behavioral: Healthy Eating Education Learning (HEAL)
  Arms: Healthy Eating Education Learning (HEAL)

SUMMARY:
PRIMARY OBJECTIVE(S):

To evaluate the efficacy of the Brief Behavioral Therapy for Insomnia (BBT-I) in treating insomnia among breast cancer patients receiving chemotherapy.

SECONDARY OBJECTIVE(S):

* To evaluate the efficacy of the BBT-I in treating cancer-related symptoms such as cancer-related fatigue and cognitive difficulties in breast cancer patients receiving chemotherapy.
* To examine potential moderators and mediators of BBT-I intervention effects on insomnia, cognitive difficulties, and fatigue. In particular, we are interested in age, depression and anxiety and side effects (hot flashes) as potential moderators of the intervention effects as well as evaluating modifiable behavioral and physiological mechanisms as hypothesized mediators

ELIGIBILITY:
INCLUSION CRITERIA

* Female
* Diagnosis of Breast Cancer (Stage I-IIIA)
* Scheduled for planned cancer treatment (eg, chemotherapy or biologic agents), or treatment is continuing
* Has ≥ 6 weeks of cancer treatment (eg, chemotherapy or biologic agents) remaining
* ≥ 21 years of age.
* Able to understand written and spoken English.
* Sleep disturbance of 8 or greater on the ISI, and insomnia that began or got worse with diagnosis of cancer or treatment with chemotherapy (to exclude pre-existing, chronic insomnia).
* Karnofsky score ≥ 70

EXCLUSION CRITERIA

* Have an unstable self-reported medical or psychiatric illness (Axis I - current or within the last 5 years).
* Be currently pregnant or nursing
* History of substance abuse or meet criteria for current alcohol abuse or dependence
* History (self-reported) of sleep apnea or restless leg syndrome (RLS)
* Self-report or have a medical record of an unstable comorbid medical or psychiatric condition that would make it unsafe or impossible to adhere to the study protocol
* Unable or unwilling to discontinue anxiolytics within 4 hours of education sessions
* Irregular heartbeat or arrhythmia (self-reported or in the medical record)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult females ≥ 21 years of age
Enrollment: 139 (Actual)
Dates: Start 2015-01; Primary Completion 2019-06-19 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oxana Palesh, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Woldeamanuel YW, Blayney DW, Jo B, Fisher SE, Benedict C, Oakley-Girvan I, Kesler SR, Palesh O. Headache outcomes of a sleep behavioral intervention in breast cancer survivors: Secondary analysis of a randomized clinical trial. Cancer. 2021 Dec 1;127(23):4492-4503. doi: 10.1002/cncr.33844. Epub 2021 Aug 6. PMID 34357593

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Eating Education Learning (HEAL): Control group. Healthy Eating Education Learning (HEAL)
- Brief Behavioral Therapy for Insomnia (BBT-I): Experimental Group. Brief Behavioral Therapy for Insomnia (BBT-I)
Period: Overall Study
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
Started | 66 | 73
Completed | 66 | 73
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I) | Total
Number analyzed (Participants) | 66 | 73 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 63 | 126
  >=65 years | 3 | 10 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (10.0) | 51.1 (11.5) | 50.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 73 | 139
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 | 20
  Not Hispanic or Latino | 48 | 62 | 110
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 15 | 32
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 2 | 4 | 6
  White | 40 | 49 | 89
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 66 | 73 | 139

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: The effects of the Brief Behavioral Therapy for Insomnia (BBT-I) intervention on insomnia will be measured by the Insomnia Severity Index (ISI). The ISI survey questionnaire is a 7-question survey, with each question having 5 possible answers (none, mild, moderate, severe, or very severe), scored as 0, 1, 2, 3, or 4, respectively. The full range of ISI scores is from 0 to 28. Lower scores are considered good, better, or healthy, and increasingly higher scores are considered to indicate greater insomnia. Clinical interpretation is as follows:
  * 0 to 7 = No clinically significant insomnia
  * 8 to14 = Sub-threshold insomnia (mild)
  * 15 to 21 = Clinical insomnia (moderate severity)
  * 22 to 28 = Clinical insomnia (severe) ISI survey will be conducted at baseline, post intervention, 6 months and 12 months. The outcome is reported as the mean ISI score at baseline; immediately post-intervention (6 weeks nominal); 6 months; and 12 months.
Time Frame: 12 months
Population: T2 (Post intervention): 5 participants were lost to follow up & didn't complete any measures.
  T3 (6 months follow-up): 16 participants did not complete any measures & were lost to follow up (including 2 deceased).
  T4 (12 months follow-up): 14 participants did not complete any measures & were lost to follow up (including 3 deceased).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
Number analyzed (Participants) | 66 | 73
score on a scale
  T1 (Baseline) | 13.73 (5.11) | 14.93 (4.84)
  T2 (Post intervention): number analyzed (Participants) | 65 | 69
  T2 (Post intervention) | 11.28 (5.43) | 10.16 (4.31)
  T3 (6 months follow-up): number analyzed (Participants) | 62 | 61
  T3 (6 months follow-up) | 9.53 (5.33) | 8.87 (5.87)
  T4 (12 months follow-up): number analyzed (Participants) | 63 | 62
  T4 (12 months follow-up) | 9.51 (5.35) | 8.98 (4.93)

2. Secondary Outcome: Brief Fatigue Inventory (BFI)
Description: The Brief Fatigue Inventory (BFI) survey questionnaire is a 9-question survey, with each question having 11 possible answers ("No fatigue" to "As bad as you can imagine"), scored from 0 to 10, with the total score being the sum of a participant's individual questions scores at a timepoint and will range from 0 to 90. Lower scores are considered good, better, or healthy, and increasingly higher scores are considered to indicate greater fatigue.
  The BFI survey was conducted at baseline, post intervention, 6 months, and 12 months. The outcome is reported as the mean of the overall BFI scores with standard deviation at baseline, immediately post-intervention (6 weeks nominal), 6 months, and 12 months.
Time Frame: 12 months
Population: T2: 5 participants were lost to follow up & did not complete any measures. T3: 16 participants did not complete any measures & were lost to follow up (including 2 deceased).
  T4: 14 participants did not complete any measures & were lost to follow up (including 3 deceased).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
Number analyzed (Participants) | 66 | 73
score on a scale
  T1 (Baseline) | 4.44 (2.28) | 4.02 (2.27)
  T2 (Post intervention): number analyzed (Participants) | 65 | 69
  T2 (Post intervention) | 4.32 (2.20) | 3.88 (2.20)
  T3 (6 months follow-up): number analyzed (Participants) | 62 | 61
  T3 (6 months follow-up) | 3.27 (2.07) | 3.00 (2.03)
  T4 (12 months follow-up): number analyzed (Participants) | 63 | 62
  T4 (12 months follow-up) | 3.28 (2.18) | 2.80 (2.09)

3. Secondary Outcome: Clinical Assessment of Depression (CAD)
Description: Anxiety and depression will be assessed by administration of the Clinical Assessment of Depression (CAD). The CAD questionnaire is a 50-item survey, with each statement having 4 possible responses ("Strongly Disagree" to "Strongly Agree"), scored from 1 to 4, The raw scores are then converted to T-scores. A score of 50 represents the mean. A difference of 10 from the mean in either the positive or negative direction indicates a difference of one standard deviation.
  The CAD survey was conducted at baseline, post intervention, 6 months, and 12 months. The outcome is reported as the mean of the overall CAD scores with standard deviation at baseline, immediately post-intervention (6 weeks nominal), 6 months, and 12 months.
Time Frame: 12 months
Population: T2(Post intervention): 6 participants were lost to follow & did not complete any measures.
  T3(6 months follow-up): 19 participants did not complete follow-up study visit & were lost to follow up (including 2 deceased).
  T4(12 months follow-up): 17 participants did not complete follow-up study visit & were lost to follow up (including 3 deceased).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
Number analyzed (Participants) | 66 | 73
score on a scale
  T1 (Baseline) | 54.38 (11.86) | 55.44 (10.80)
  T2 (Post intervention): number analyzed (Participants) | 64 | 69
  T2 (Post intervention) | 53.14 (11.25) | 54.32 (11.59)
  T3 (6 months follow-up): number analyzed (Participants) | 60 | 60
  T3 (6 months follow-up) | 51.15 (13.13) | 51.40 (10.58)
  T4 (12 months follow-up): number analyzed (Participants) | 62 | 60
  T4 (12 months follow-up) | 49.74 (12.58) | 50.60 (10.66)

4. Secondary Outcome: Comprehensive Trail Making Test (CTMT)
Description: Neuropsychological assessments will be conducted using the Comprehensive Trail Making Test (CTMT), an assessment of simple attention and executive function, consisting of 5 dot-to-dot exercises that increase with complexity and difficulty. A score of 50 represents the mean. A difference of 10 from the mean in either the positive or negative direction indicates a difference of one standard deviation. Thus, a score of 60 is one standard deviation above the mean, while a score of 30 is two standard deviations below the mean. Overall, higher values indicate better executive functioning, attention, and processing speed.
  The CTMT assessment was conducted at baseline, post intervention, 6 months, and 12 months. The outcome is reported as the mean of the overall CTMT scores with standard deviation at baseline, immediately post-intervention (6 weeks nominal), 6 months, and 12 months.
Time Frame: At baseline, post intervention, 6 months and 12 months
Population: T1(Baseline): 1 participant did not complete baseline assessment. T2(Post intervention): Total 7 participants were not analyzed; 6 participants were lost to follow up and 1 participant did not complete this measure T3(6 months follow-up): 19 participants did not complete follow-up (including 2 deceased).
  T4(12 months follow-up): 18 participants did not complete follow-up(including 3 deceased).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
Number analyzed (Participants) | 66 | 73
score on a scale
  T1 (Baseline): number analyzed (Participants) | 65 | 73
  T1 (Baseline) | 44.22 (7.76) | 41.44 (7.98)
  T2 (Post intervention): number analyzed (Participants) | 63 | 69
  T2 (Post intervention) | 48.68 (8.79) | 45.04 (8.68)
  T3 (6 months follow-up): number analyzed (Participants) | 60 | 60
  T3 (6 months follow-up) | 48.68 (8.29) | 46.53 (8.33)
  T4 (12 months follow-up): number analyzed (Participants) | 61 | 60
  T4 (12 months follow-up) | 49.26 (7.86) | 47.92 (7.56)

5. Secondary Outcome: Hopkins Verbal Learning Test Revised (HVLT-R) Sub-test for Delayed Recall
Description: Neuropsychological assessments will be conducted using the Delayed Recall sub-test from the overall Hopkins Verbal Learning Test Revised (HVLT-R). The result values are known as the T score. A higher T scores indicating better memory (recall).A score of 50 represents the mean. A difference of 10 from the mean in either the positive or negative direction indicates a difference of one standard deviation
  The HVLT-R sub-test assessment for Delayed Recall was conducted at baseline, post intervention, 6 months, and 12 months. The outcome is reported as the mean score with standard deviation at baseline, immediately post-intervention (6 weeks nominal), 6 months, and 12 months.
Time Frame: At baseline, post intervention, 6 months and 12 months
Population: T2 (Post intervention): 6 participants were lost to follow up & did not complete any measures.
  T3(6 months follow-up): 18 participants did not complete follow-up study visit (including 2 deceased).
  T4(12 months follow-up): 17 participants did not complete follow-up study visit (including 3 deceased).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
Number analyzed (Participants) | 66 | 73
score on a scale
  T1 (Baseline) | 49.05 (10.83) | 49.42 (9.58)
  T2 (Post intervention): number analyzed (Participants) | 64 | 69
  T2 (Post intervention) | 49.06 (10.95) | 46.96 (11.05)
  T3 (6 months follow-up): number analyzed (Participants) | 61 | 60
  T3 (6 months follow-up) | 50.70 (9.78) | 51.68 (9.63)
  T4 (12 months follow-up): number analyzed (Participants) | 62 | 60
  T4 (12 months follow-up) | 52.95 (8.30) | 52.68 (8.67)

6. Secondary Outcome: Hopkins Verbal Learning Test Revised (HVLT-R) Sub-test for Verbal Learning & Memory
Description: Neuropsychological assessments will be conducted using the Verbal Learning and Memory sub-test from the overall Hopkins Verbal Learning Test Revised (HVLT-R). The result values are known as the T score.The higher T scores indicating better memory (recall). A score of 50 represents the mean. A difference of 10 from the mean in either the positive or negative direction indicates a difference of one standard deviation
  The HVLT-R sub-test assessment for Verbal Learning and Memory was conducted at baseline, post intervention, 6 months, and 12 months. The outcome is reported as the mean score with standard deviation at baseline, immediately post-intervention (6 weeks nominal), 6 months, and 12 months.
Time Frame: At baseline, post intervention, 6 months and 12 months
Population: T2(Post intervention): 6 participants were lost to follow up & did not complete any measures.
  T3 (6 months follow-up): 18 participants did not complete follow-up visit (including 2 deceased).
  T4 (12 months follow-up): 17 participants did not complete follow-up visit (including 3 deceased).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
Number analyzed (Participants) | 66 | 73
score on a scale
  T1 (Baseline) | 48.94 (11.45) | 50.23 (11.30)
  T2 (Post intervention): number analyzed (Participants) | 64 | 69
  T2 (Post intervention) | 49.44 (12.27) | 50.42 (11.32)
  T3 (6 months follow-up): number analyzed (Participants) | 61 | 60
  T3 (6 months follow-up) | 53.21 (10.78) | 53.85 (9.66)
  T4 (12 months follow-up): number analyzed (Participants) | 62 | 60
  T4 (12 months follow-up) | 56.05 (9.60) | 56.93 (9.99)

7. Secondary Outcome: Controlled Oral Word Association Test (COWAT)
Description: Neuropsychological assessments will be conducted using the Controlled Oral Word Association Test (COWAT), a verbal fluency task that assesses complex cognition. The test value is the the count of words that meet pre-defined criteria within 1 minute, so the minimum is 0 and no fixed maximum exists. Adjustments are made to the raw score based on participant age and education level, resulting in a scaled score. Higher scores reflect a better outcome, meaning better cognition and verbal fluency.
  The COWAT assessment was conducted at baseline, post intervention, 6 months, and 12 months. The outcome is reported as the mean of the COWAT score with standard deviation at baseline, immediately post-intervention (6 weeks nominal), 6 months, and 12 months.
Time Frame: At baseline, post intervention, 6 months and 12 months
Population: T2: 6 participants were lost to follow & did not complete any measures. T3: 18 participants did not complete the 6-month follow-up study visit & were lost to follow up (including 2 deceased).
  T4: 17 participants did not complete the 12-month follow-up study visit & were lost to follow up (including 3 deceased).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
Number analyzed (Participants) | 66 | 73
score on a scale
  T1 (Baseline) | 41.95 (9.87) | 39.51 (11.97)
  T2 (Post intervention): number analyzed (Participants) | 64 | 69
  T2 (Post intervention) | 42.19 (11.36) | 40.43 (12.36)
  T3 (6 months follow-up): number analyzed (Participants) | 61 | 60
  T3 (6 months follow-up) | 45.72 (11.11) | 43.53 (12.06)
  T4 (12 months follow-up): number analyzed (Participants) | 62 | 60
  T4 (12 months follow-up) | 44.61 (10.22) | 42.73 (11.77)

8. Secondary Outcome: Mobile Cognitive Assessment Battery (MCAB)
Description: Cognitive difficulties will be assessed by administration of the Mobile Cognitive Assessment Battery (MCAB), comprised of 3 neuropsychological tests and a self-reported assessment. MCAB measures cognitive flexibility, accuracy, processing speed, working memory and multitasking.
  The MCAB survey was to be conducted at baseline, post intervention, 6 months, and 12 months. The outcome was to be reported as the mean of the overall MCAB scores with standard deviation at baseline, immediately post-intervention (6 weeks nominal), 6 months, and 12 months.
Time Frame: At baseline, post intervention, 6 months and 12 months
Population: No analysis. The MCAB analysis was determined to not be a validated measure, and the analysis was not conducted as the scores are not standardized and results do not have meaning at this time.
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 52 months
Arm/Group | Healthy Eating Education Learning (HEAL) | Brief Behavioral Therapy for Insomnia (BBT-I)
All-Cause Mortality (participants affected / at risk) | 0/66 | 3/73
Serious Adverse Events (participants affected / at risk) | 3/66 | 7/73
Other Adverse Events (participants affected / at risk) | 17/66 | 19/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Eating Education Learning (HEAL) (N=66) | Brief Behavioral Therapy for Insomnia (BBT-I) (N=73)
Disease Progression (General disorders) | 0 (0) | 3 (3)
Blood Transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Eating Education Learning (HEAL) (N=66) | Brief Behavioral Therapy for Insomnia (BBT-I) (N=73)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Infection: not specified (Infections and infestations) | 2 (2) | 1 (1)
Allergic reaction (Immune system disorders) | 4 (5) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Breast infection (Infections and infestations) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 3 (3) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify:Dermatomyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain- cardiac (Cardiac disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders- other, specify: Crohn's (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Infusion related reaction: GI symptoms (unspecified) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Localized Edema (General disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intraoperative breast injury: Breast necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT02165839/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT02165839/Prot_SAP_001.pdf